CLINICAL TRIAL: NCT03840707
Title: LIFEwithIBD: Living With Intention, Fullness and Engagement With Inflammatory Bowel Disease: The Impact of a Group Intervention and an ICT-based Transcultural Intervention on Physical and Mental Health
Brief Title: LIFEwithIBD: Living With Intention, Fullness and Engagement With Inflammatory Bowel Disease
Acronym: LIFEwithIBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, Inês A Trindade, Dr, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUC-068-18
Record Dates: First submitted 2019-02-05; First posted 2019-02-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): LIFEwithIBD Programme is a manualized acceptance, mindfulness and compassionate-based group intervention for inflammatory bowel disease patients. It included 9 weekly group sessions, 1.30h hours each, run in small groups (ranging from 10 to 15 participants).
  Participants in this group also receive inflammatory bowel disease treatment as usually performed at the Coimbra University Hospital.
  Interventions: Behavioral: LIFEwithIBD
- Control group (No Intervention): Treatment as Usual (TAU) Standard personalized treatment of inflammatory bowel disease

INTERVENTIONS:
Behavioral: LIFEwithIBD — LIFEwithIBD programme is a psychotherapeutic programme based on Acceptance, Mindfulness and Compassion for inflammatory bowel disease patients
  Treatment as Usual (TAU): Standard personalized treatment of inflammatory bowel disease
  Arms: Experimental group

SUMMARY:
This investigation aims to apply and test the feasibility of an acceptance, mindfulness and compassionate-based intervention structured for inflammatory bowel disease patients. LIFEwithIBD programme for inflammatory bowel disease thus comprises 9 weekly group sessions, lasting 1 and a half hour each, run in small groups at a Gastroenterology Service at the Coimbra's University Hospital. For each week participants have assigned homework (e.g., mindfulness exercises). The efficacy of LIFE-IBD Group Intervention to improve quality of life, mental health, and disease activity-related scores will be tested in a sample of Portuguese patients. Additionally, this study expected that the observable changes after the intervention completion will be attributed to changes in emotional regulation processes and maintained over the follow-up periods.

DETAILED DESCRIPTION:
The sample will include diagnosed inflammatory bowel disease patients recruited at a Gastroenterology Service at the Coimbra's University Hospital, a national reference centre for IBD. Patients will be approached by their doctor to assess their level of interest in the investigation. Patients who demonstrate interest will go through a Screening interview conducted by a psychologist that aims explain the structure and arms of the investigation, to collect demographic data, and whether the patient meets the inclusion criteria for the study. After sample collection, participants will be randomly assigned to one of two conditions: experimental group (n=75) or control group (n=75). The experimental group will be divided into five subgroups of 15 participants. The first group will function as a pilot group to test the suitability of the programme. The intervention will include 8 weekly sessions, with the duration of 90 minutes each. Groups will have two therapists with experience in ACT and CFT-based interventions. All participants will continue on receiving the recommended pharmacological treatment for IBD (TAU). This will allow the comparison between the participants receiving the LIFE-IBD Group Intervention+TAU (experimental group) and the participants only receiving TAU (control group). The frequency of engagement with the programme at home practises will be analysed as moderator of the efficacy of the programme. Both groups will concurrently complete a protocol of measures to assess main three areas: a) psychological processes; b) quality of life and psychopathology; c) current medical status. These assessments will occur in four different times: before the start of the LIFEwithIBD programme M0), after the final session of the programme (M1), and 3 (M2) and 6 months (M4) after that.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of IBD for more than 6 months (CD or UC)

Exclusion Criteria:

* having started new treatment for IBD in the previous 6 months (in the case of anti-TNF and immunosuppressive therapy) or 2 months (in the case of steroid or aminosalicylate therapy)
* cognitive impairment;
* currently undergoing any form of psychological intervention;
* current diagnosis of severe psychiatric illness (severe depression, psychotic illness, bipolar disorder, substance abuse) or suicidal ideation;
* diagnosis of other serious health condition;
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Indicators of psychopathology (DASS-21) | From Baseline to 3-months follow-up
  Indicators of psychopathology, namely depression, anxiety and stress symptoms will be measured by Depression, Anxiety and Stress Scale-21. DASS-21 assesses levels of depression, anxiety, and stress symptoms. Respondents are asked to indicate how frequently they experienced such symptoms over the previous week on a 4-point scale (ranging from 0 = "Did not apply to me at all" to 3 = "Applied to me very much, or most of the time"). Results of each subscale are calculated by the sum of the results of the seven items. The scale provides three notes, one per subscale, where the minimum is "0" and the maximum is "21". Higher results correspond to more negative affective states.

SECONDARY OUTCOMES:
Perception of Quality of Life (World Health Organization Brief Quality of Life Assessment Scale) | From Baseline to 3-months follow-up
  Quality of life will be measure by World Health Organization Brief Quality of Life Assessment Scale.The WHOQOL-BREF is a 24-item measure of subjective perceptions of QoL. Items are rated on a 5-point Likert scale (higher scores indicate perceptions of higher QoL) and are distributed over four domains-physical health (e.g. "To what extent do you feel that physical pain prevents you from doing what you need to do?"), psychological health (e.g. "How often do you have negative feelings such as blue mood, despair, anxiety, depression?"-reverse item),social relationships (e.g. "How satisfied are you with your personal relationships?"), and environment. The scale also presents two additional items that evaluate general quality of life and general health.
Biochemical indicator: concentration levels of calprotectin | From Baseline to 3-months follow-up
  This biochemical indicator will be measured though concentration levels of calprotectin in unit of measure of miligram/liter (mg/L)
Biochemical indicator: concentration levels of C-reactive protein (CRP) | From Baseline to 3-months follow-up
  This biochemical indicator will be measured though concentration levels of C-reactive protein (CRP) in unit of measure of microgram/gram (µg/g)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

REFERENCES:
- [Derived] Ferreira C, Pereira J, Skvarc D, Oliveira S, Galhardo A, Ferreira NB, Lucena-Santos P, Carvalho SA, Matos-Pina I, Rocha BS, Portela F, Trindade IA. Randomized controlled trial of an Acceptance and Commitment Therapy and compassion-based group intervention for persons with inflammatory bowel disease: the LIFEwithIBD intervention. Front Psychol. 2024 May 9;15:1367913. doi: 10.3389/fpsyg.2024.1367913. eCollection 2024. PMID 38784617
- [Derived] Trindade IA, Pereira J, Galhardo A, Ferreira NB, Lucena-Santos P, Carvalho SA, Oliveira S, Skvarc D, Rocha BS, Portela F, Ferreira C. The LIFEwithIBD Intervention: Study Protocol for a Randomized Controlled Trial of a Face-to-Face Acceptance and Commitment Therapy and Compassion-Based Intervention Tailored to People With Inflammatory Bowel Disease. Front Psychiatry. 2021 Aug 19;12:699367. doi: 10.3389/fpsyt.2021.699367. eCollection 2021. PMID 34489756